CLINICAL TRIAL: NCT02418091
Title: STOP-DKD Automated Population Program (APP)
Brief Title: Integrated Population Program for Diabetic Kidney Disease
Acronym: STOP-DKD APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00052081; 1R34DK102166-01 (NIH)
Record Dates: First submitted 2015-03-20; First posted 2015-04-16 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Diabetic Kidney Disease; Uncontrolled Hypertension
Keywords: patients with moderate DKD and uncontrolled HTN
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Telehealth (Experimental): Using Telehealth to slow progression of diabetic kidney disease automated population program identifies patients and engages them to optimize DKD medication adherence and health behaviors using 2-way communication via patient-selected technology (mobile/web-based applications, text messaging, interactive voice response, or e-mail) backed by case management via the phone for suboptimal control or health status. The STOP-DKDAutomated Population Program will deliver a tailored, multi-factorial intervention to address medication self-management and modify multiple risk factors simultaneously through a combination of patient self-monitoring, behavioral therapies and education that optimize adherence and self-efficacy.
  Interventions: Behavioral: Telehealth
- Control/No Intervention (No Intervention): Group of subjects that will serve as a comparison group. These subjects will not be approached/enrolled for this study.

INTERVENTIONS:
Behavioral: Telehealth — Using Telehealth to slow progression of diabetic kidney disease automated population program identifies patients and engages them to optimize DKD medication adherence and health behaviors using 2-way communication via patient-selected technology (mobile/web-based applications, text messaging, interactive voice response, or e-mail) backed by case management via the phone for suboptimal control or health status. The STOP-DKDAutomated Population Program will deliver a tailored, multi-factorial intervention to address medication self-management and modify multiple risk factors simultaneously through a combination of patient self-monitoring, behavioral therapies and education that optimize adherence and self-efficacy.
  Arms: Intervention Telehealth

SUMMARY:
This study will build a population management system Simultaneous risk factor control using Telehealth to slOw Progression of Diabetic Kidney Disease STOP-DKD Application STOP-DKD APP and conduct a 6-month controlled trial to compare reduction of blood pressure. In addition, the study will evaluate the feasibility of future large-scale intervention to slow diabetic kidney disease (DKD) DKD progression.

Aim 1: Identify patients with moderate DKD and uncontrolled hypertension (HTN) using existing electronic health record data in an integrated data warehouse (Southeastern Diabetes Initiative- SEDI) to screen all patients within SEDI.

Aim 2: Implement an intervention designed to slow progression of DKD and treat associated conditions in a high-risk population with moderate DKD and uncontrolled HTN using the STOP-DKD APP

* Primary Outcome: Test the hypothesis that patients who receive the intervention will have greater improvements in blood pressure as compared to a control group after 6 months
* Secondary Outcomes: Exploratory analyses to determine whether patients who receive the intervention will have less progression (defined as a smaller decrease in kidney function), and improved behaviors that affect HTN control and cardiovascular risk (medication adherence, diet, physical activity, and weight control) as compared to a control group after 6 months

Aim 3: Evaluate the STOP-DKD APP Study to guide large-scale implementation & dissemination

* Impact Evaluation: Assess the potential population impact of our intervention using the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework
* Economic Evaluation: Conduct an economic evaluation using the Archimedes Model by estimating projected costs and quality-adjusted life-years

ELIGIBILITY:
Potentially eligible patients will be identified using the existing SEDI (Southeastern Diabetes Initiative) data warehouse that pulls electronic health record data quarterly from ten different source systems in the four counties.

* Adults (age ≥18 and 75 years);
* Diagnosis of type 2 diabetes (ICD-9 codes 250.x0, 250.x2);
* Have at least 2 serum creatinine values available in the 3 prior years, separated by at least 3 months;
* Preserved kidney function (based upon the last year's eGFR average of between 45-90 ml/min/1.73m2, estimated by calculating an eGFR using the 4-variable Modification of Diet in Renal Disease study equation);
* Evidence of diabetic nephropathy (Either: 1. presence of macroalbuminuria; 2. history of microalbuminuria prior to ACE (angiotensin-converting enzyme) inhibitor or angiotensin receptor blocker (ARB) therapy; 3. previous documentation of diabetic retinopathy or laser therapy; 4. if only microalbuminuria and no #3, then urinalysis without hematuria, and no other renal etiologies [i.e., glomerulonephritis, polycystic kidney disease, membranous nephropathy, renal artery stenosis])
* Uncontrolled HTN (1y mean clinic SBP≥140 and/or DBP≥90).

Exclusion Criteria:

Patients who meet any one of the exclusion criteria will be excluded:

* No access to telephone
* Not proficient in English
* Nursing home/long-term care facility resident or receiving home health care
* Impaired hearing/ speech/ vision
* Participating in another trial (pharmaceutical or behavioral)
* Planning to leave the area in the next 3 years
* Pancreatic insufficiency or diabetes secondary to pancreatitis
* Alcohol abuse (>14 alcoholic beverages/ wk)
* Diagnosis of non-diabetic kidney disease
* Active malignancy (other than non-melanomatous skin cancer)
* Diagnosis of life-threatening disease with death probable within 4 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure | Baseline & 6months

SECONDARY OUTCOMES:
Change in estimated Glomerular filtration rate (eGFR) for kidney function | Baseline & 6months
Change in dietary habits as measured by questionnaire | Baseline & 6month
Change in weight | Baseline & 6month
Change in amount of physical activity as measured by questionnaire | Baseline & 6month
  Investigators will assess whether patients who receive the intervention will have improved behaviors that affect HTN control and cardiovascular risk ( physical activity) as compared to a control group after 6 months
Change in taking medicine as prescribed | Baseline& 6month
  Investigators will assess whether patients who receive the intervention will have improved behaviors that affect HTN control and cardiovascular risk (medication adherence) as compared to a control group after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Uptal Patel, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] Lewinski AA, Patel UD, Diamantidis CJ, Oakes M, Baloch K, Crowley MJ, Wilson J, Pendergast J, Biola H, Boulware LE, Bosworth HB. Addressing Diabetes and Poorly Controlled Hypertension: Pragmatic mHealth Self-Management Intervention. J Med Internet Res. 2019 Apr 9;21(4):e12541. doi: 10.2196/12541. PMID 30964439